CLINICAL TRIAL: NCT00463450
Title: A Multicenter, Double-blind, Randomized, Cross-over Study to Investigate the Efficacy of Gynodian® Depot i.m. Compared to 4 mg Estradiol Valerate i.m. Both Given Every Four Weeks for Five Months Combined With 5 mg Medroxyprogesterone Acetate Orally in Postmeno-pausal Women With Impaired Well-being, Mood and Sexuality
Brief Title: Efficacy of Gynodian® Depot in Women With Impaired Well-being
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Navitas Life Sciences GmbH (Industry); LKF Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 90651; 303401
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Hormone Replacement Therapy
Keywords: Hormone Replacement Therapy; Impaired well-being, mood and sexuality
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Gynodian® Depot (BAY86-5032)
- Arm 2 (Active Comparator)
  Interventions: Drug: BAY86-4980

INTERVENTIONS:
Drug: Gynodian® Depot (BAY86-5032) — Injection monthly
  Arms: Arm 1
Drug: BAY86-4980 — orally
  Arms: Arm 2

SUMMARY:
The typical menopausal symptoms that are associated with a variety of physical and psychological changes (e.g. nervousness, anxiety, and depression) and also with impaired sexual interest and enjoyment are caused by a lack of estrogen, a female sex hormone produced inside the body. To treat these symptoms, women who are postmenopausal can receive a therapy called 'hormone replacement therapy' (the dosage of hormones to replace the body's deficient hormones), for instance, with estrogen preparations injected into a muscle.In women with a uterus estrogen use causes the lining of the womb (endometrium) to grow (thicken) as before the menopause. With long-term use this may lead to pathological changes of the endometrium. That is why this therapy should be complemented by the estrogens' natural counterbalance, progesterone (progestogen), at a certain interval. This causes the lining of the womb to shed, with monthly bleeding like a normal period, thus avoiding excessive endometrial growth.Estrogen treatment is well known to relieve psychological complaints. The combination of an estrogen with a weak androgen (in this case Dehydroepiandrosterone (DHEA)) is presumed to clearly increase this effect. The present clinical study is to prove that Gynodian? Depot as a combination of estrogen and androgen has a better effect on psychological complaints and sexuality in postmenopausal women than has treatment with the estrogen Estradiol valerate alone.All patients will receive the same therapy, but differing in sequence. Either they receive Gynodian? Depot during the first five cycles and the estrogen-only preparation during cycles 6-10 (treatment group 1) or they receive the study medication in reverse order (treatment group 2). Patients will be assigned to one of the two groups at random. In either case they will be given an injection into the gluteal muscle every four weeks.Women with an intact uterus, in addition to the injections (the day of the injection being the 1st day of a cycle) have to take a tablet containing 5 mg Medroxyprogesterone acetate (MPA) (progestogen) per day for 14 days (cycle days 15-28) to enable the endometrium to shed in a monthly period.The study will extend over a total period of about 11 months, during which the patient will have 16 appointments for examinations.After patient has signed on the informed consent form for participation in this clinical study, the investigator will ask her, which diseases she has at the moment or has had during the past 12 months and which medicinal products she has been taking. Subsequently, she will have a gynecological examination (including the breasts) as well as a general physical examination. Blood pressure, heart rate as well as body height and weight will be measured and noted down. In addition, the doctor will question her about physical and psychological menopausal complaints by means of two different, short questionnaires. Only if the evaluation of these two questionnaires shows that she is eligible for the participation in this clinical study, will the following actions be carried through.Approx. 40 ml blood will be taken from the patient for a thorough laboratory test including her hormone levels, and she will be asked for a urine sample. Additionally, she will have a vaginal ultrasound examination of the womb lining, a cervical smear test (unless already done during the last three months), and an x-ray examination of the breasts (mammography) (unless already done during the last 12 months).These measures will be repeated at Final visit.About 3 weeks after visit 1, when the investigator has the results of all tests prescribed at visit 1, the patient will be asked to appear for visit 2.If the patient is eligible for a participation in this clinical study, she will be given the first injection of the study medication.During the following visits, injections will be given, blood pressure and pulse rate as well as body weight will be measured and blood will be drawn to measure the hormone levels.All procedures will apply also during the second treatment period. When switching to the second treatment period a physical and gynecological examination will additionally be performed.Questionnaires have to be filled in by the patient at different time points during the study.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Postmenopausal status (amenorrhea for at least 12 months)
* 45 - 65 years of age
* Application of estrogen or cyclic estrogen/progestin preparation other than the study medication for at least 6 months prior to Visit 1
* Relevant impairment of well-being and mood inspite of estrogen therapy (confirmed by questionnaire scores)
* BMI<33kg/m2

Exclusion Criteria:

* Uterine bleeding of unknown etiology within the last 2 years
* Previous or existing or suspected carcinoma of the breast
* Any malignant disease in the last 5 years
* Endometrial double layer thickness > 5 mm
* History of thromboembolic events or existing thromboembolic processes
* Prior hormone replacement therapy with androgens within 12 months prior to Visit 1
* Major life events within the last 12 months prior to Visit 1

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2002-05; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
To assess the difference in the Global Severity Index (GSI) of both treatment sequences with Gynodian Depot and with estradiol valerate | After 4.5 cycles of treatment

SECONDARY OUTCOMES:
To assess the difference in the GSI in both treatment sequences | After 1.5 cycles of treatment
To assess the difference in the scores of the psychometric tests and rating scales SCL-90-R, Menopause rating scale, HADS and Visual analog Scale in both treatment sequences | After 1.5 and 4.5 cycles of treatment
To assess serum hormone levels of DHEA, DHEAS, androsterone, testosterone, dihydrotestosterone, androstenediol-glucuronid, estradiol, estrone, and SHBG | At end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer